CLINICAL TRIAL: NCT04672161
Title: Education Intervention on Vaccination Adherence Among IBD Patients at Weill Cornell Medical Center
Brief Title: Education Intervention on Vaccination Adherence Among Inflammatory Bowel Disease (IBD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-06022242
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Crohn Disease (CD); Ulcerative Colitis (UC); Indeterminate Colitis
Keywords: Vaccine; HPV; Vaccination; IBD; Inflammatory Bowel Diseases; UC; CD
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine Education (Experimental): Patients randomized to the Experimental arm will receive a baseline educational intervention on vaccination following a vaccination history survey. Patients will be followed 6-months after the intervention to record prospective clinical data. Evidence of vaccination-status will be documented. Besides standard of care visits and testing, no additional procedures will be carried out for the purpose of this study.
  Interventions: Other: Vaccine Education
- No Vaccine Education (No Intervention): Patients randomized to the No Intervention arm will not receive the Vaccine Education. They will only complete the survey on their vaccination history.

INTERVENTIONS:
Other: Vaccine Education — A baseline educational intervention on vaccination and its role in the health maintenance of patients with IBD will be provided to all participants. Those on immunosuppressive therapies and/or those age 65 or older will also be offered the pneumonia vaccine educational intervention. Finally, patients aged 18-26 and those 27-45 who have never been vaccinated for HPV or those with high risk for HPV will additionally receive the HPV educational intervention.
  Arms: Vaccine Education

SUMMARY:
A retrospective chart review and a six-month prospective outcome analysis aimed to evaluate the efficacy of a vaccination education intervention and vaccination adherence among IBD patients at Weill-Cornell Medical Center. It is hypothesized that a general vaccination education campaign will improve vaccination adherence rates for all IBD patients. Secondarily, it is hypothesized that an Human Papilloma Virus (HPV) vaccination intervention targeted at high-risk IBD patients will increase vaccination adherence among these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Weill-Cornell Medical Center with an in-person or virtual appointment between March 1 - August 30, 2021.
* Documentation of an IBD diagnosis (CD, UC, IC).

Exclusion Criteria:

* No documentation of an IBD diagnosis.
* Pregnant or breastfeeding.
* No scheduled appointment between March 1-August 30, 2021.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Mean Change in Vaccination Adherence in Patients | Baseline; 6 months

SECONDARY OUTCOMES:
Change in qualitative attitude assessment on vaccination adherence and non-adherence as measured by self-reported 6-month questionnaire. | Baseline; 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dana J Lukin, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No